CLINICAL TRIAL: NCT01386879
Title: Evaluation of Microaspiration and Efficacy of Above the Cuff Suctioning During General Anesthesia: A Comparison of Two Endotracheal Tubes With Suction Above Cuff With a Standard Endotracheal Tube
Brief Title: Evaluation of Above the Cuff Suctioning During General Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated because of slower than anticipated enrollment
Sponsor: Thomas Jefferson University (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11D.48
Record Dates: First submitted 2011-06-27; First posted 2011-07-01 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Secretion Removal Above ETT Cuff
Keywords: suction; aspiration; general anesthesia; intubation; endotracheal tube; respiratory complications
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- TaperGuard Evac ETT (Experimental): Trachea will be intubated with Mallinckrodt™TaperGuard™ Evac Endotracheal Tube with a suction port to facilitate removal of secretions from the region of the trachea below the vocal cords and above the inflated ETT cuff
  Interventions: Drug: methylene blue
- Teleflex ISIS ETT (Experimental): Trachea will be intubated with Teleflex ISIS HVT Cuffed Tracheal Tube with Subglottic Secretion suction port to facilitate removal of secretions from the region of the trachea below the vocal cords and above the inflated ETT cuff
  Interventions: Drug: methylene blue
- Standard ETT (Active Comparator): Control group of patients will be intubated with a standard ETT without a suction port above the cuff (The Mallinckrodt Intermediate Hi-Lo Endotracheal Tube)
  Interventions: Drug: methylene blue

INTERVENTIONS:
Drug: methylene blue — A dilute solution of methylene blue (5 ml of 1 % methylene blue solution in saline, 1:1 dilution) will be gently delivered into the hypopharynx using a flexible suction catheter approximately once per hour until trachea is extubated.
  Other Names: Urolene Blue

SUMMARY:
The aim of this prospective, randomized, pilot study is compare ease of tracheal intubation, amount of microaspiration and efficacy of secretion removal using three FDA (Food and Drug Administration)-cleared endotracheal tubes (ETT) after the induction of general anesthesia in the operating room (OR). Studies in the intensive care unit (ICU) have demonstrated a significant reduction in the incidence of ventilator acquired pneumonia when a ETT with suction above the cuff is used to remove secretions that accumulate above the inflated cuff. This will be the first study to evaluate the efficacy of above the cuff suctioning during general anesthesia and surgery.

One hundred and ten adult patients undergoing elective abdominal surgery (general, colorectal or gynecological) requiring general anesthesia with an endotracheal tube and mechanical ventilation will be randomized into 3 groups to receive one of the following three endotracheal tubes:

1. Teleflex ISIS HVT Cuffed Tracheal Tube with Subglottic Secretion Suction Port Endotracheal Tube (Teleflex ISIS ETT).
2. Mallinckrodt TaperGuard Evac Endotracheal Tube (TaperGuard Evac ETT).
3. Mallinckrodt Intermediate Hi-Lo Endotracheal Tube. (Standard ETT)

The first two groups will be compared to standard ETT (third group) regarding easy of tracheal intubation, efficacy of suctioning of secretions, efficacy of sealing the trachea with an inflated ETT cuff by preventing the movement of test dye (methylene blue) from the pharynx into the trachea and incidence of post-operative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective abdominal surgery with an anticipated duration longer than 2 hours.
* ASA (American Society of Anesthesiologists) Physical status Classification 1 to 3. (1 - normal healthy patient, 2 - patients with mild systemic disease, 3 - patients with severe systemic disease)
* Endotracheal intubation anticipated to be routine (not difficult) based upon preoperative airway assessment

Exclusion Criteria:

* Short duration surgery (anticipated < 2 hours) or emergency (non-elective) surgery
* ASA Physical status Classification 4 to 5. (4 - patients with severe systemic diseases that is a constant threat to life, 5 - Moribund patients who are not expected to survive without the operation)
* Anticipated difficult airway requiring technique other than direct laryngoscopy for intubation of the trachea.
* Pregnancy
* History of allergic reaction to Methylene Blue medication
* Methemoglobinemia, glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of symptomatic chronic obstructive pulmonary disease (asthma, bronchitis, emphysema) or recent pneumonia (< 6 months prior to surgery).
* Hypoxemia (hemoglobin oxygen saturation < 90% room air or on O2 at home or in hospital)
* History of coagulopathy, IV heparin therapy, or coumadin therapy (INR > 2.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We did initial 10 roll-in subjects to be familiar with all of the procedures and recordings.
Period: Overall Study
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT
Started | 17 | 17 | 16
Completed | 17 | 17 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT | Total
Number analyzed (Participants) | 17 | 17 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.88 (8.62) | 55.53 (15.00) | 54.56 (12.85) | 54.66 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 22
  Male | 10 | 10 | 8 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 28.40 (3.25) | 26.23 (4.12) | 26.85 (4.41) | 27.16 (3.92)
ASA [Count of Participants; unit: Participants] — American Society of Anesthesiology Physical Status:
  ASA I: A normal healthy patient. ASA II: A patient with mild systemic disease. ASA III: A patient with a severe systemic disease that is not life-threatening
  Participants
    I | 0 | 2 | 2 | 4
    II | 12 | 9 | 8 | 29
    III | 5 | 6 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Prevention of the Movement of Test Dye (Methylene Blue) From the Pharynx Into Patients' Trachea During Surgery
Description: The primary objective of the pilot study is to evaluate whether there is a difference between the 3 types of ETT in preventing the movement of test dye (methylene blue) from the pharynx into the trachea, past the inflated cuff. After tracheal intubation a small amount of methylene blue will be instilled into patients' pharynx every 60 minutes. The presence or absence of blue dye above and below the ETT cuff will be evaluated every 20 minutes using a video recording fiberoptic bronchoscope.
Time Frame: 4 hours
Population: the number of participants with dye in the distal trachea. One bronchoscopy recording was corrupted and not able to be evaluated in the GEvac group.
Measure: Number; unit: number of participants with dye
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT
Number analyzed (Participants) | 16 | 17 | 16
number of participants with dye | 0 | 0 | 2

2. Secondary Outcome: Evaluation of pH of Secretions Collected Above Endotracheal Tube Cuff During Surgery
Description: Secretions will be continuously suctioned from the suction port of the two ETT with suction above the cuff port (TaperGard Evac ETT and Teleflex ISIS ETT) into a Luken's trap. We will evaluate whether there is a difference in the pH of the aspirate between two ETT with suction above the cuff port.
Time Frame: 4 hours
Population: Average Secretion pH
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT
Number analyzed (Participants) | 17 | 17
pH | 7.38 (0.59) | 7.29 (0.41)

3. Secondary Outcome: the Ease of Tracheal Intubation Following the Induction of General Anesthesia Among the 3 Types of ETT
Description: Time to intubate trachea
Time Frame: 1 hour
Population: Time to intubate trachea in all groups
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT
Number analyzed (Participants) | 17 | 17 | 16
minutes | 7.53 (0.48) | 7.59 (0.48) | 7.41 (0.58)

4. Secondary Outcome: Evaluation the Trachea and Vocal Cords at the Time of ETT Extubation to Determine Whether There is a Difference in the Amount of Mucosal Injury Between the 3 Types of ETT.
Description: number of patients with mucosal injury and blood below the vocal cords
Time Frame: 4 hours
Population: Extubation bronchoscopy data. some data are not available in all groups
Measure: Count of Participants; unit: Participants
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT
Number analyzed (Participants) | 13 | 16 | 14
Participants | 10 | 11 | 7

5. Secondary Outcome: Evaluation of Volume of Secretions Collected Above Endotracheal Tube Cuff During Surgery
Description: Secretions will be continuously suctioned from the suction port of the two ETT with suction above the cuff port (TaperGard Evac ETT and Teleflex ISIS ETT) into a Luken's trap.
Time Frame: 4 hours
Population: Total Secretion Volume collected in Luken's trap. NO data for standard groups since there was no suction port in the standard ETT
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT
Number analyzed (Participants) | 17 | 17
mL | 13.00 (10.48) | 26.00 (19.01)

6. Secondary Outcome: Evaluation of Bacterial Load of Secretions Collected Above Endotracheal Tube Cuff During Surgery
Description: Secretions will be continuously suctioned from the suction port of the two ETT with suction above the cuff port (TaperGard Evac ETT and Teleflex ISIS ETT) into a Luken's trap. The number of patients with a bacterial load of the aspirate between two ETT with suction above the cuff port was measured by gram stain of the aspirated secretions.
Time Frame: 4 hours
Population: Only two groups that had suction above the cuff had the collected secretions and were analyzed. The specimen was Gram Stained and the presence of any bacteria/organisms was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT
Number analyzed (Participants) | 17 | 17
Participants | 13 | 13

ADVERSE EVENTS:
Time Frame: 24 h
Description: Postoperative pulmonary complications (pneumonia, aspiration pneumonitis, atelectasis, pleural effusion or respiratory insufficiency/failure).
Arm/Group | TaperGuard Evac ETT | Teleflex ISIS ETT | Standard ETT
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 1/17 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TaperGuard Evac ETT (N=17) | Teleflex ISIS ETT (N=17) | Standard ETT (N=16)
post-operative cough, sputum production or wheezing within 24 hours (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) — post-operative cough, sputum production or wheezing within 24 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No